CLINICAL TRIAL: NCT00712751
Title: The Sexual Health of Rectal Cancer Patients: a Pilot Study
Brief Title: The Sexual Health of Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Albert Einstein College of Medicine (Other); Icahn School of Medicine at Mount Sinai (Other); M.D. Anderson Cancer Center (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-073
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer; Rectum
Keywords: Rectum; Quality of Life; Sexual Health; 08-073
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: usual care (UC) which is the standard care that patients receive
  Interventions: Behavioral: questionnaires
- 2: Cancer Survivorship Intervention-Sexual Health (CSI-SH)plus Usual Care (US)
  Interventions: Behavioral: CSI-SH- Cancer Survivorship Intervention

INTERVENTIONS:
Behavioral: questionnaires — Participants randomized to the Usual Care arm will receive standard care . For women, this is defined as the care that participants who are not in the intervention receive; we will ask these participants what psychosocial care they are receiving to track usual care. For men, "usual care" will consist of a standardized referral to the men's Sexual Medicine Program at MSKCC and written information in the form of the American Cancer Society (ACS) booklet on Sexuality after Cancer. Individuals randomized to Usual Care will not receive any additional counseling sessions from the study interventionists until they are done with the follow up interviews and then it will be offered to them. Follow up questionnaires will assess all study participants at 4 and 8 months after baseline.
  Groups: 1
Behavioral: CSI-SH- Cancer Survivorship Intervention — This involves four 1-hour individual sessions with three additional telephone booster/review sessions provided in between the four sessions. Sessions can be completed in person or conducted over the phone. Although every effort will be made to complete the booster session in between counseling sessions, if the patient is unavailable to complete the booster calls they may be skipped. Sessions one and two will focus on rehabilitation techniques and tools will be provided and discussed with participants during these first two sessions.
  Groups: 2

SUMMARY:
We know that treatment for rectal, colorectal or anal cancer can impact sexual function. This study aims to learn:

* How the treatment affects emotional and social well-being.
* How a new sexual health educational program affects you.

Cancer patients seek education for lots of reasons. It often helps them cope because they can express their feelings with a trained professional. This study is open to individuals who have been treated for rectal, colorectal or anal cancer. It involves a new type of sexual health counseling program. It will teach participants skills that they can use to improve their sex lives. These skills may also improve physical and emotional well-being. We will compare the new type of sexual health program with the standard care patients receive after treatment for rectal, colorectal or anal cancer.

DETAILED DESCRIPTION:
This is a two year randomized clinical trial examining the feasibility, tolerability, acceptability (including adherence) and efficacy of an intervention designed to improve sexual functioning of survivors of rectal cancer.

We have completed enrollment of female patients and are currently collecting follow up data. Recruitment for male patients is ongoing. Male participants will now be randomized in a 3:1 ratio to either the intervention condition (n = 40) or the control condition (n = 40).

ELIGIBILITY:
Inclusion Criteria:

* At least six months post radiation and/or surgery for stage I-III rectal adenocarcinoma or rectosigmoid for cancer with an anastomosis at 15 cm or below and completed treatment
* At least six months post radiation and/or chemotherapy for anal cancer.
* Have no evidence of disease or recurrence
* For women indicate Indicate moderate satisfaction or below on their overall sexual life (a score of "4" or lower on the question "Over the past 4 weeks, how satisfied have you been with your overall sexual life?"
* For men indicate, and a score of "3" or lower on the question "How would you rate your confidence that you could get and keep an erection" for men) and a score of "2" or higher on the question "How much does this problem bother you?
* In the judgment of the consenting professional interventionists, able to communicate in English well enough to work with English speaking and complete the study assessments.
* Age 21 years or older.

Exclusion Criteria:

* Significant cognitive or psychiatric disturbance sufficient, in the investigator's judgment, to preclude participation in a psychotherapeutic intervention.
* Are actively participating in protocol 06-151
* Participated in focus group or qualitative interview.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal patients
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2008-06-24 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
To investigate the feasibility, tolerability, acceptability (including adherence) and efficacy of CSI-SH, a psycho-educational intervention, on the primary outcome of sexual functioning among RC survivors. | conclusion of study

SECONDARY OUTCOMES:
To investigate the impact of CSI-SH on secondary outcomes: sexual self-schema, cancer specific distress, general distress symptoms, and Quality of Life for all participants, as well as sexual bother for men only. | conclusion of study
To explore baseline variables that may influence the effectiveness of CSI-SH (i.e., moderators such as socio-demographic and medical variables). | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Nelson CJ, Schuler TA, Reiner AS, Baser RE, Demirjian CC, Mulhall J, Temple L, Schover L, Jandorf L, DuHamel KN. A psychoeducational intervention to improve sexual functioning in male rectal and anal cancer patients: A pilot randomized controlled trial study. Palliat Support Care. 2024 Feb 23:1-9. doi: 10.1017/S1478951523001906. Online ahead of print. PMID 38389458
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org